CLINICAL TRIAL: NCT01341158
Title: Neoadjuvant Treatment of Locoregional Metastases in Malignant Melanoma (AJCC Stage IIIB/C) With Multiferon: a Phase IIa DeCOG Trial
Brief Title: NAM-Trial: Multiferon in Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Benjamin Weide, M.D., Dr. Benjamin Weide, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5021000
Record Dates: First submitted 2011-04-19; First posted 2011-04-25 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Locoregional Metastases in Malignant Melanoma Stages IIIB/C
Keywords: Malignatn Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Drug: human interferon-α

INTERVENTIONS:
Drug: human interferon-α — Neoadjuvant treatment: Multiferon is given as flat dosages (3 - 9 - 18 MIU) 5 days per week, subcutaneously for 4 weeks
  Other Names: Multiferon

SUMMARY:
The current clinical trial shall clarify the efficacy, safety and biologic effects of neoadjuvant treatment with natural interferon-α (Multiferon) in patients with locoregional metastases of melanoma in stage IIIB/C.

DETAILED DESCRIPTION:
The study is an open label, multicenter phase IIa clinical trial which is designed as a pilot project in order to establish the efficacy and tolerability of Multiferon as a neoadjuvant treatment of locoregional metastases. Patients will be treated subsequently in cohorts characterized by different doses (3 - 9 - 18 MIU) to analyze dosage dependent effects.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven cutaneous melanoma
2. Clinical stage IIIB or IIIC (AJCC 2010)
3. ≥ 18 years of age
4. Presence of at least two metastases, not more than 10 metastases, and completely resectable
5. Measurable disease (at least one lesion that can be accurately measured in two perpendicular diameters, with both dimensions at least 10 mm x 10 mm for spiral CT and 5 mm x 5 mm for locoregional metastases assessed by ultrasound or digital photography)
6. ECOG performance status of 0/1
7. Patients with previous adjuvant recombinant interferon-α treatment of any dose are eligible if (i) treatment was stopped at least 1 month before start of treatment and (ii) no progression occurred during interferon-α treatment.
8. No childbearing potential or negative pregnancy test within 14 days before inclusion in women with child bearing potential Women with childbearing potential must be using an effective method of contraception (Pearl-Index < 1, e.g. oral contraceptives, other hormonal contraceptives [vaginal products, skin patches, or implanted or injectable products], or mechanical products such as an intrauterine device or barrier methods [diaphragm, spermicides]) throughout the study and for up to 3 months after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.

   No men of fathering potential or men of fathering potential must be using an effective method of contraception to avoid conception throughout the study and for up to 3 months after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.
9. Signed and dated informed consent informed consent before the start of specific protocol procedures

Exclusion Criteria:

1. Mucous membrane or ocular melanoma
2. Any evidence of distant metastasis (e.g. whole body CT-scan including brain scan within 4 weeks before inclusion)
3. Patients with severe cardiac disease (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months before inclusion, ventricular tachyarrhythmia requiring ongoing treatment, unstable angina pectoris).
4. ALAT or ASAT > 2 x ULN
5. Total bilirubin > 2 x ULN
6. Creatinine > 2 x ULN
7. Evidence or history of depression. If this condition can not be ruled out, the patient should be transferred to a psychiatrist for consultation and further assessment before inclusion.
8. Patients with seizure disorders requiring anticonvulsant therapy
9. Any of the following abnormal baseline hematologic/laboratory values:

   Hb < 10g/dl WBC < 3.0x109 /l Platelets < 100x109 /l
10. Presence of active autoimmune disease
11. Concurrent systemic glucocorticoids or any other systemic immunosuppressive therapy
12. Unwilling or unable to comply with the requirements of the protocol
13. Known infection with HBV, HCV, HIV
14. Pregnant or lactating women
15. Unwillingness or inability to employ an effective barrier method of birth control throughout the study and for up to 3 months after end of treatment in female or male patients
16. Known or suspected allergy to human interferon alpha or any ingredient of the IMP.
17. Any thyroid dysfunctions not responsive to therapy
18. Presence of chronic hepatitis with decompensated liver cirrhosis
19. Immunosuppression in patients with transplantation
20. Evidence or history of bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | after 4 weeks of treatment
  Overall response rate (clinical and radiological) after 4 weeks of treatment (CR + PR) according to immune-related response criteria (irRC)

SECONDARY OUTCOMES:
Disease control rate | after 4 weeks of treatment
  Disease control rate (CR + PR +SD) according to irRC
Rate of histopathological complete responses | after 4 weeks of treatment
  Rate of histopathological complete responses
Tolerability | after 4 weeks of treatment
  Assessment of numbers of adverse events
Differences in gene expression in metastatic tissue before/after treatment | after 4 weeks of treatment
Dose dependency of effects | after 4 weeks of treatment
Changes of serum markers and PBMC subsets before/after treatment (optional translational side studies) | after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätshautklinik Tübingen, Tübingen, Germany